CLINICAL TRIAL: NCT04622709
Title: Pilot Study of Loop Diuretics Among Individuals Receiving Hemodialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-3550; 1R03DK124651-01 (NIH)
Record Dates: First submitted 2020-10-02; First posted 2020-11-10 (Actual); Results first posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hemodialysis; Dialysis; End Stage Renal Disease; Patient-reported Outcomes; Symptoms; Diuretic; Furosemide; Lasix
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Furosemide; Sodium Potassium Chloride Symporter Inhibitors; Tablets

STUDY DESIGN:
Intervention Model Description: This is a single-center (multi-clinic), open-label, non-randomized pilot study to test whether oral furosemide is safe and effective at increasing urine volume in HD patients. The study will consist of 2 periods: a 6-week dose escalation period (period 1) and a subsequent 12-week follow-up period (period 2). During period 1, all participants will receive escalating doses of furosemide as tolerated, and the short-term safety, tolerability, and efficacy of furosemide will be examined. During period 2, all participants will continue the maximally tolerated period 1 furosemide dose, and the acceptability of and adherence to furosemide and the longer-term safety and efficacy of furosemide will be examined.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study drug administration: furosemide (Experimental): Study participants will receive furosemide oral tablets to be taken twice daily. During study period 1 (first 6 weeks), the drug dose will be escalated every 2 weeks if safe, tolerated, and acceptable to the participant. During study period 2 (subsequent 12 weeks), participants will take the maximum tolerated dose from study period 1, received every 4 weeks if safe, tolerated, and acceptable to the participant.
  Interventions: Drug: Furosemide (loop diuretic) Tablets

INTERVENTIONS:
Drug: Furosemide (loop diuretic) Tablets — Open label dose escalation study of furosemide in people receiving maintenance hemodialysis. Participants will take furosemide oral tablets twice daily for 18 weeks. Doses will be titrated every 2 weeks for 6 weeks if safe, effective, tolerated, and accepted by the participant. First 2 weeks of the study: participants not taking oral furosemide at enrollment will take 80mg furosemide twice daily, those taking oral furosemide at enrollment will stay on their prescribed dose, and those taking another loop diuretic at enrollment will discontinue their prescription and take an equivalent oral furosemide dose. At week 4: dose escalation if tolerated (from 80mg to 120mg twice daily for the 1st group, and a 50% increased dose not >320mg/day for the 2nd & 3rd groups). At week 6: dose escalation if tolerated (from 120mg to 160mg twice daily for the 1st group, and a 50% increased dose not >320mg/day for the 2nd & 3rd groups). Final 12 weeks: all participants will take the maximum tolerated dose.

SUMMARY:
Individuals with kidney failure receiving maintenance hemodialysis (HD) have high mortality rates, driven largely by cardiovascular causes. Volume-related factors are critical, modifiable contributors to cardiovascular complications. Reversing volume overload has been shown to improve blood pressure and cardiac remodeling. Use of loop diuretics may represent a pragmatic, low-cost, and low-burden strategy to improve outcomes in people receiving HD. Lack of data on optimal furosemide dosing, safety, and acceptability are barriers to expanded use. This study investigates whether oral furosemide is safe and effective at increasing urine volume in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient self-report of at least 1 cup urine/24-hours
* Age ≥18 years
* Receipt of thrice weekly in-center HD at a participating clinic (UNC-associated Carolina Dialysis- Carrboro, Siler City, Pittsboro, Sanford, and Lee County)
* ≥60 days receiving in-center HD
* Willingness to take study medication and undergo study testing
* Ability to provide informed consent

Exclusion Criteria:

* Known allergy to loop diuretic
* History of poor adherence to HD or medical regimen per nephrologist
* >1 hospitalization in prior 30-days
* Frequent hypotension (systolic BP <80 mmHg at >30% of HD treatments in prior 30-days)
* Cirrhosis per nephrologist
* Hearing disorder per nephrologist
* Serum potassium <3.5 mEq/L, magnesium <1 mg/dL, or corrected calcium <8 mg/dL in prior 30-days
* Taking a non-loop diuretic (e.g. spironolactone, eplerenone, ethacrynic acid, thiazides)
* Taking an aminoglycoside, cisplatin, methotrexate, cyclosporine, adrenocorticotropic hormone (ACTH), lithium, phenytoin, or oral/intravenous steroid
* Natural licorice consumption
* Prisoners, patients with significant mental illness
* Pregnant patients and nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Flythe, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - Carolina Dialysis - Carrboro, Carrboro, North Carolina
  - Carolina Dialysis - Pittsboro, Pittsboro, North Carolina
  - Carolina Dialysis - Sanford, Sanford, North Carolina
  - Carolina Dialysis - Lee County, Sanford, North Carolina
  - Carolina Dialysis - Siler City, Siler City, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data that supports the results will be shared from 9 through 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From 9 months through 36 months after publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug Administration: Furosemide: Open label dose escalation study of furosemide in people receiving maintenance hemodialysis. Participants will take furosemide oral tablets twice daily for 18 weeks. This was a single-arm study with 2 periods. Period 1 is the dose escalation phase. During period 1 (first 6 weeks), the drug dose will be escalated every 2 weeks if safe, tolerated, and acceptable to the participant. Period 2 is the follow-up phase. During period 2 (subsequent 12 weeks), all participants will take the maximum tolerated dose from study period 1, received every 4 weeks if safe, tolerated, and acceptable to the participant.
  First 2 weeks of the study: participants not taking oral furosemide at enrollment will take 80mg furosemide twice daily, those taking oral furosemide at enrollment will stay on their prescribed dose, and those taking another loop diuretic at enrollment will discontinue their prescription and take an equivalent oral furosemide dose. At week 4: dose escalation if tolerated (from 80mg to 120mg twice daily for the 1st group, and a 50% increased dose not >320mg/day for the 2nd & 3rd groups). At week 6: dose escalation if tolerated (from 120mg to 160mg twice daily for the 1st group, and a 50% increased dose not >320mg/day for the 2nd & 3rd groups). Final 12 weeks: all participants will take the maximum tolerated dose (period 2).
  In this single-arm study, all participants received oral furosemide. The protocol was pre-specified to summarize outcome events as a single arm.
Period: Period 1 (First 6 Weeks)
Arm/Group | Study Drug Administration: Furosemide
Started | 39
Completed | 36
Not Completed | 3
Period: Period 2 (Subsequent 12 Weeks)
Arm/Group | Study Drug Administration: Furosemide
Started | 36
Completed | 32
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [58 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have a Defined Increase in 24-hour Urine Volume From Baseline to Week 5
Description: Participants will follow standard dialysis clinic protocols for 24-urine volume collection. Classifying participants as has having an increase in 24-hour urine volume will be contingent on the amount of urine the participant makes at baseline.
  * Among participants with baseline 24-hour urine volume ≥200 mL: ≥25% increase in urine volume is considered an increase.
  * Among participants with baseline 24-hour urine volume <200 mL: ≥50 mL increase in urine volume to a urine volume of at least 100 mL/24-hours is considered an increase.
  The percentage of participants who have a defined increase in 24-urine volume from baseline to week 5 will be determined.
Time Frame: Baseline and study week 5 (5 weeks after study medication start
Population: Summarizing outcome events as a single arm (i.e., patients with a baseline 24-hour urine volume ≥200 mL and < 200 mL as a single group) was pre-specified in the protocol. 36 participants completed the week 5 24-hour urine volume collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
percentage of participants | 33

2. Primary Outcome: Percentage of Participants Who Have a Defined Increase in 24-hour Urine Volume From Baseline to Week 12
Description: Participants will follow standard dialysis clinic protocols for 24-urine volume collection. Classifying participants as has having an increase in 24-hour urine volume will be contingent on the amount of urine the participant makes at baseline.
  * Among participants with baseline 24-hour urine volume ≥200 mL: ≥25% increase in urine volume is considered an increase.
  * Among participants with baseline 24-hour urine volume <200 mL: ≥50 mL increase in urine volume to a urine volume of at least 100 mL/24-hours is considered an increase.
  The percentage of participants who have a defined increase in 24-urine volume from baseline to week 12 will be determined.
Time Frame: Baseline and study week 12 (12 weeks after study medication start)
Population: Summarizing outcome events as a single arm (i.e., patients with a baseline 24-hour urine volume ≥200 mL and < 200 mL as a single group) was pre-specified in the protocol. 33 participants completed the week 12 24-hour urine volume collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 33

3. Primary Outcome: Percentage of Participants Who Have a Defined Increase in 24-hour Urine Volume From Baseline to Week 18
Description: Participants will follow standard dialysis clinic protocols for 24-urine volume collection. Classifying participants as has having an increase in 24-hour urine volume will be contingent on the amount of urine the participant makes at baseline.
  * Among participants with baseline 24-hour urine volume ≥200 mL: ≥25% increase in urine volume is considered an increase.
  * Among participants with baseline 24-hour urine volume <200 mL: ≥50 mL increase in urine volume to a urine volume of at least 100 mL/24-hours is considered an increase.
  The percentage of participants who have a defined increase in 24-urine volume from baseline to week 18 will be determined.
Time Frame: Baseline and study week 18 (18 weeks after study medication start)
Population: Summarizing outcome events as a single arm (i.e., patients with a baseline 24-hour urine volume ≥200 mL and < 200 mL as a single group) was pre-specified in the protocol. Out of the 33 participants still enrolled in the study at week 18, 32 completed the week 18 24-hour urine volume collection. Thus, the analysis population is 32 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 32
Percentage of participants | 22

4. Primary Outcome: Percentage of Participants With A Serum Potassium <3.2 mEq/L at Week 1
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 1 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Population: 38 participants completed the week 1 blood collection. Thus, the analysis population is 38 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
percentage of participants | 0

5. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 2
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 2 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

6. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 3
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 3 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

7. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 4
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 4 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 37 participants completed the week 4 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

8. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 5
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 5 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

9. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 6
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 6 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

10. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 9
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 9 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 9 (9 weeks after study medication start)
Population: 36 participants completed the week 9 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

11. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 13
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 13 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 13 (13 weeks after study medication start)
Population: 33 participants completed the week 13 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

12. Primary Outcome: Percentage of Participants With a Serum Potassium <3.2 mEq/L at Week 17
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 17 study visit. The percentage of participants who have a serum potassium <3.2 mEq/L will be determined.
Time Frame: Study week 17 (17 weeks after study medication start)
Population: 33 participants completed the week 17 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

13. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 1
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 1 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Population: 38 participants completed the week 1 blood collection. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

14. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 2
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 2 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

15. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 3
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 3 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 blood collection. However, there was laboratory error and serum magnesium levels were only available for 36 participants. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

16. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 4
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 4 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 37 participants completed the week 4 blood collection. However, there was laboratory error and serum magnesium levels were only available for 36 participants. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

17. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 5
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 5 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

18. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 6
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 6 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

19. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 9
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 9 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 9 (9 weeks after study medication start)
Population: 36 participants completed the week 9 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

20. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 13
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 13 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 13 (13 weeks after study medication start)
Population: 33 participants completed the week 13 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

21. Primary Outcome: Percentage of Participants With a Serum Magnesium <0.8 mEq/L at Week 17
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 17 study visit. The percentage of participants who have a serum magnesium <0.8 mEq/L will be determined.
Time Frame: Study week 17 (17 weeks after study medication start)
Population: 33 participants completed the week 17 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

22. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 1
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 1 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Population: 38 participants completed the week 1 blood collection. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

23. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 2
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 2 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

24. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 3
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 3 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

25. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 4
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 4 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 37 participants completed the week 4 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

26. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 5
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 5 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

27. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 6
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 6 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

28. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 9
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 9 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 9 (9 weeks after study medication start)
Population: 36 participants completed the week 9 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

29. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 13
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 13 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 13 (13 weeks after study medication start)
Population: 33 participants completed the week 13 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

30. Primary Outcome: Percentage of Participants With a Serum Corrected Calcium <7.0 mg/dL at Week 17
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 17 study visit. The percentage of participants who have a serum corrected calcium <7.0 mg/dL will be determined.
Time Frame: Study week 17 (17 weeks after study medication start)
Population: 33 participants completed the week 17 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

31. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 1.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 1 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Population: 38 participants completed the week 1 blood collection. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

32. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 2.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 2 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

33. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 3.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 3 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

34. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 4.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 4 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 37 participants completed the week 4 blood collection. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

35. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 5.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 5 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

36. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 6.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 6 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

37. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 9.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 9 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 9 (9 weeks after study medication start)
Population: 36 participants completed the week 9 blood collection. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

38. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 13.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 13 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 13 (13 weeks after study medication start)
Population: 33 participants completed the week 13 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

39. Primary Outcome: Percentage of Participants With a Serum Furosemide Level >12 Micrograms/L at Week 17.
Description: Blood samples will be collected from participants prior to their dialysis treatments at the week 17 study visit. The percentage of participants who have a serum furosemide level >12 micrograms/L will be determined.
Time Frame: Study week 17 (17 weeks after study medication start)
Population: 33 participants completed the week 17 blood collection. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

40. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 1
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 1 will be determined.
Time Frame: Up to study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 0

41. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 2
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 2 will be determined.
Time Frame: Up to study week 2 (2 weeks after study medication start)
Population: 38 participants were still enrolled in the study at week 2. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

42. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 3
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 3 will be determined.
Time Frame: Up to study week 3 (3 weeks after study medication start)
Population: 38 participants were still enrolled in the study at week 3. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

43. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 4
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 4 will be determined.
Time Frame: Up to study week 4 (4 weeks after study medication start)
Population: 38 participants were still enrolled in the study at week 4. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

44. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 5
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 5 will be determined.
Time Frame: Up to study week 5 (5 weeks after study medication start)
Population: 36 participants were still enrolled in the study at week 5. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

45. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 6
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 6 will be determined.
Time Frame: Up to study week 6 (6 weeks after study medication start)
Population: 36 participants were still enrolled in the study at week 6. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

46. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 7
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 7 will be determined.
Time Frame: Up to study week 7 (7 weeks after study medication start)
Population: 36 participants were still enrolled in the study at week 7. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

47. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 8
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 8 will be determined.
Time Frame: Up to study week 8 (8 weeks after study medication start)
Population: 36 participants were still enrolled in the study at week 8. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

48. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 9
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 9 will be determined.
Time Frame: Up to study week 9 (9 weeks after study medication start)
Population: 36 participants were still enrolled in the study at week 9. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

49. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 10
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 10 will be determined.
Time Frame: Up to study week 10 (10 weeks after study medication start)
Population: 36 participants were still enrolled in the study at week 10. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

50. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 11
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 11 will be determined.
Time Frame: Up to study week 11 (11 weeks after study medication start)
Population: 34 participants were still enrolled in the study at week 11. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

51. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 12
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 12 will be determined.
Time Frame: Up to study week 12 (12 weeks after study medication start)
Population: 34 participants were still enrolled in the study at week 12. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

52. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 13
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 13 will be determined.
Time Frame: Up to study week 13 (13 weeks after study medication start)
Population: 34 participants were still enrolled in the study at week 13. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

53. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 14
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 14 will be determined.
Time Frame: Up to study week 14 (14 weeks after study medication start)
Population: 34 participants were still enrolled in the study at week 14. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

54. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 15
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 15 will be determined.
Time Frame: Up to study week 15 (15 weeks after study medication start)
Population: 34 participants were still enrolled in the study at week 15. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

55. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 16
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 16 will be determined.
Time Frame: Up to study week 16 (16 weeks after study medication start)
Population: 34 participants were still enrolled in the study at week 16. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

56. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 17
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 17 will be determined.
Time Frame: Up to study week 17 (17 weeks after study medication start)
Population: 33 participants were still enrolled in the study at week 17. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

57. Primary Outcome: Percentage of Participants That Experience Dialysis-associated Hypotension up to Week 18
Description: Participants' blood pressure will be measured with an upper extremity cuff in a seated position at 15-minute intervals during each hemodialysis treatment per standard dialysis clinic protocols. Dialysis-associated hypotension will be defined as hypotension during dialysis requiring hospitalization or treatment in an emergency room and not attributable to overt sepsis, acute myocardial infarction, or other cardiovascular event (e.g. aortic dissection). The percentage of participants who have dialysis-associated hypotension up to week 18 will be determined.
Time Frame: Up to study week 18 (18 weeks after study medication start)
Population: 33 participants were still enrolled in the study at week 18. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

58. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 0

59. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

60. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

61. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

62. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

63. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

64. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

65. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

66. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

67. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

68. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

69. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Rash Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious rash will be defined as rash ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe rash attributable to furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

70. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 0

71. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

72. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 3

73. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 3

74. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 3

75. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 3

76. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 3

77. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

78. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 3

79. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

80. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

81. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Tinnitus Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious tinnitus will be defined as tinnitus ranked as severe or very severe and attributable to furosemide. Incidence will be defined as percentage of participants who have serious tinnitus. The percentage of participants reporting severe or very severe tinnitus attributable to furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

82. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 0

83. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

84. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

85. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

86. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

87. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

88. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

89. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

90. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

91. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

92. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

93. Primary Outcome: Percentage of Participants Reporting a Severe or Very Severe Hearing Change Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious hearing change will be defined as hearing change ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting a severe or very severe hearing change attributable to furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

94. Primary Outcome: Change in the Inner EAR Instrument Score From Baseline to Week 1
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 1. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score.
Time Frame: Baseline and study week 1 (1 week after study medication start)
Population: This outcome was entered in error. Data was not collected on this outcome, per the study protocol.
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 0

95. Primary Outcome: Percentage of Participants With a Defined Decrease in the Inner EAR Instrument Score From Baseline to Week 2
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 2. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score. The percentage of participants with a defined decrease in the Inner EAR instrument score will be determined.
Time Frame: Baseline and study week 2 (2 weeks after study medication start)
Population: 37 participants completed the Inner EAR questionnaire at week 2. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

96. Primary Outcome: Change in the Inner EAR Instrument Score From Baseline to Week 3
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 3. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score.
Time Frame: Baseline and study week 3 (3 weeks after study medication start)
Population: This outcome was entered in error. Data was not collected on this outcome, per the study protocol.
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 0

97. Primary Outcome: Percentage of Participants With a Defined Decrease in the Inner EAR Instrument Score From Baseline to Week 4
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 4. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score. The percentage of participants with a defined decrease in the Inner EAR instrument score will be determined.
Time Frame: Baseline and study week 4 (4 weeks after study medication start)
Population: 38 participants completed the Inner EAR questionnaire at week 4. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 3

98. Primary Outcome: Change in the Inner EAR Instrument Score From Baseline to Week 5
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 5. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score.
Time Frame: Baseline and study week 5 (5 weeks after study medication start)
Population: This outcome was entered in error. Data was not collected on this outcome, per the study protocol.
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 0

99. Primary Outcome: Percentage of Participants With a Defined Decrease in the Inner EAR Instrument Score From Baseline to Week 6
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 6. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score. The percentage of participants with a defined decrease in the Inner EAR instrument score will be determined.
Time Frame: Baseline and study week 6 (6 weeks after study medication start)
Population: 36 participants completed the Inner EAR questionnaire at week 6. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

100. Primary Outcome: Change in the Inner EAR Instrument Score From Baseline to Week 8
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 8. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score.
Time Frame: Baseline and study week 8 (8 weeks after study medication start)
Population: This outcome was entered in error. Data was not collected on this outcome, per the study protocol.
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 0

101. Primary Outcome: Percentage of Participants With a Defined Decrease in the Inner EAR Instrument Score From Baseline to Week 10
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 10. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score. The percentage of participants with a defined decrease in the Inner EAR instrument score will be determined.
Time Frame: Baseline and study week 10 (10 weeks after study medication start)
Population: 36 participants completed the Inner EAR questionnaire at week 10. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

102. Primary Outcome: Change in the Inner EAR Instrument Score From Baseline to Week 12
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 12. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score.
Time Frame: Baseline and study week 12 (12 weeks after study medication start)
Population: This outcome was entered in error. Data was not collected on this outcome, per the study protocol.
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 0

103. Primary Outcome: Percentage of Participants With a Defined Decrease in the Inner EAR Instrument Score From Baseline to Week 14
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 14. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score. The percentage of participants with a defined decrease in the Inner EAR instrument score will be determined.
Time Frame: Baseline and study week 14 (14 weeks after study medication start)
Population: 33 participants completed the Inner EAR questionnaire at week 14. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

104. Primary Outcome: Change in the Inner EAR Instrument Score From Baseline to Week 16
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 16. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score.
Time Frame: Baseline and study week 16 (16 weeks after study medication start)
Population: This outcome was entered in error. Data was not collected on this outcome, per the study protocol.
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 0

105. Primary Outcome: Percentage of Participants With a Defined Decrease in the Inner EAR Instrument Score From Baseline to Week 18
Description: Participants' hearing ability during the last week will be assessed using the Inner Effectiveness of Auditory Rehabilitation (Inner EAR) 11-question validated questionnaire administered during study week 18. The total instrument score will be tallied at each administration [range: 10 (low hearing ability) - 59 (high hearing ability)]. Serious hearing change will be defined as a ≥10-point decrease in the Inner EAR instrument score from baseline score. The percentage of participants with a defined decrease in the Inner EAR instrument score will be determined.
Time Frame: Baseline and study week 18 (18 weeks after study medication start)
Population: 33 participants completed the Inner EAR questionnaire at week 18. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 6

106. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 10

107. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 16

108. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 11

109. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 11

110. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 17

111. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 6

112. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 8

113. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 17

114. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 12

115. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 9

116. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 6

117. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Cramping Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious cramping will be defined as cramping ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe cramping attributable to furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 9

118. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 3

119. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 5

120. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

121. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 3

122. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 6

123. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

124. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

125. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

126. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 3

127. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

128. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

129. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Dizziness/Pre-syncope Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious dizziness/pre-syncope will be defined as dizziness/pre-syncope ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe dizziness/pre-syncope attributable to furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

130. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 0

131. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

132. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

133. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

134. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

135. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

136. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

137. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

138. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 3

139. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 6

140. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

141. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Unusual Tiredness/Weakness Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the prior week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious unusual tiredness/weakness will be defined as unusual tiredness/weakness ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe unusual tiredness/weakness will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

142. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 0

143. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

144. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

145. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

146. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

147. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

148. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

149. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

150. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 0

151. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

152. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

153. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Chest Pain Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious chest pain will be defined as chest pain ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe chest pain will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

154. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 5

155. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

156. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 3

157. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 3

158. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 8

159. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

160. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 6

161. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

162. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 6

163. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

164. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

165. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Nausea Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious nausea will be defined as nausea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe nausea will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

166. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 3

167. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

168. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

169. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

170. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

171. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

172. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

173. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

174. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 3

175. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 6

176. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

177. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Vomiting Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious vomiting will be defined as vomiting ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe vomiting will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 3

178. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 1
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 1. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 39
Percentage of participants | 3

179. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 2
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 2. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 37 participants completed the week 2 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

180. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 3
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 3. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 37 participants completed the week 3 symptom questionnaire. Thus, the analysis population is 37 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 37
Percentage of participants | 0

181. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 4
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 4. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 38 participants completed the week 4 symptom questionnaire. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 0

182. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 5
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 5. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 36 participants completed the week 5 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

183. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 6
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 6. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 36 participants completed the week 6 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

184. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 8
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 8. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 36 participants completed the week 8 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 3

185. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 10
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 10. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 36 participants completed the week 10 symptom questionnaire. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 0

186. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 12
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 12. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 34 participants completed the week 12 symptom questionnaire. Thus, the analysis population is 34 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 34
Percentage of participants | 6

187. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 14
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 14. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 33 participants completed the week 14 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 6

188. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 16
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 16. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 33 participants completed the week 16 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

189. Primary Outcome: Percentage of Participants Reporting Severe or Very Severe Diarrhea Attributable to Furosemide at Week 18
Description: Participants' dialysis-related symptoms during the last week will be assessed using an investigator-developed 13-question symptom questionnaire administered at study week 18. Each symptom will be graded using a 5-point symptom severity Likert scale (response options: none, mild, moderate, severe, very severe). Serious diarrhea will be defined as diarrhea ranked as severe or very severe and attributable to furosemide. The percentage of participants reporting severe or very severe diarrhea will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 33 participants completed the week 18 symptom questionnaire. Thus, the analysis population is 33 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 33
Percentage of participants | 0

190. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 1
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 1. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Population: 38 participants completed the week 1 acceptance assessment. Thus, the analysis population is 38 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 38
Percentage of participants | 97

191. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 2
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 2. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: 35 participants completed the week 2 acceptance assessment. Thus, the analysis population is 35 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 35
Percentage of participants | 97

192. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 3
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 3. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 35 participants completed the week 3 acceptance assessment. Thus, the analysis population is 35 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 35
Percentage of participants | 94

193. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 4
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 4. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: Out of the 38 participants still enrolled in the study at week 4, 32 participants completed the week 4 adherence assessment. Thus, the analysis population is 32 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 32
Percentage of participants | 94

194. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 5
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 5. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 31 participants completed the week 5 acceptance assessment. Thus, the analysis population is 31 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 31
Percentage of participants | 90

195. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 6
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 6. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 31 participants completed the week 6 acceptance assessment. Thus, the analysis population is 31 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 31
Percentage of participants | 97

196. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 8
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 8. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 31 participants completed the week 8 acceptance assessment. Thus, the analysis population is 31 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 31
Percentage of participants | 90

197. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 10
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 10. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 28 participants completed the week 10 acceptance assessment. Thus, the analysis population is 28 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 28
Percentage of participants | 89

198. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 12
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 12. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 26 participants completed the week 12 acceptance assessment. Thus, the analysis population is 26 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 26
Percentage of participants | 96

199. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 14
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 14. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 26 participants completed the week 14 acceptance assessment. Thus, the analysis population is 26 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 26
Percentage of participants | 96

200. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 16
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 16. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 26 participants completed the week 16 acceptance assessment. Thus, the analysis population is 26 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 26
Percentage of participants | 96

201. Primary Outcome: Percentage of Participants Reporting Acceptance of Furosemide at Week 18
Description: Participants' acceptance of furosemide will be assessed using an investigator-developed 1-question questionnaire administered at study week 18. Patient-reported acceptance of furosemide at the dose during which the questionnaire is administered will be defined as an affirmative response ("yes") to the question "If recommended, would you be willing to stay on the dose of furosemide you have received during the last week?". The percentage of participants reporting acceptance of furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 25 participants completed the week 18 acceptance assessment. Thus, the analysis population is 25 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 25
Percentage of participants | 92

202. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 1
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 1. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 1 (1 week after study medication start)
Population: 36 participants completed the week 1 pill counts. Thus, the analysis population is 36 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 36
Percentage of participants | 67

203. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 2
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 2. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 2 (2 weeks after study medication start)
Population: Out of the 38 participants still enrolled in the study at week 2, 32 participants completed the week 2 pill counts. Thus, the analysis population is 32 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 32
Percentage of participants | 81

204. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 3
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 3. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 3 (3 weeks after study medication start)
Population: 21 participants completed the week 3 pill counts. Thus, the analysis population is 21 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 21
Percentage of participants | 52

205. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 4
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 4. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 4 (4 weeks after study medication start)
Population: 30 participants completed the week 4 pill counts. Thus, the analysis population is 30 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 30
Percentage of participants | 67

206. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 5
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 5. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 5 (5 weeks after study medication start)
Population: 27 participants completed the week 5 pill counts. Thus, the analysis population is 27 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 27
Percentage of participants | 81

207. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 6
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 6. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 6 (6 weeks after study medication start)
Population: 26 participants completed the week 6 pill counts. Thus, the analysis population is 26 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 26
Percentage of participants | 81

208. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 8
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 8. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 8 (8 weeks after study medication start)
Population: 24 participants completed the week 8 pill counts. Thus, the analysis population is 24 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 24
Percentage of participants | 67

209. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 10
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 10. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 10 (10 weeks after study medication start)
Population: 24 participants completed the week 10 pill counts. Thus, the analysis population is 24 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 24
Percentage of participants | 75

210. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 12
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 12. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 12 (12 weeks after study medication start)
Population: 24 participants completed the week 12 pill counts. Thus, the analysis population is 24 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 24
Percentage of participants | 83

211. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 14
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 14. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 14 (14 weeks after study medication start)
Population: 25 participants completed the week 14 pill counts. Thus, the analysis population is 25 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 25
Percentage of participants | 84

212. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 16
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 16. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 16 (16 weeks after study medication start)
Population: 25 participants completed the week 16 pill counts. Thus, the analysis population is 25 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 25
Percentage of participants | 48

213. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 18
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 18. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 18 (18 weeks after study medication start)
Population: 24 participants completed the week 18 pill counts. Thus, the analysis population is 24 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 24
Percentage of participants | 75

214. Primary Outcome: Percentage of Participants Who Are Adherent to Furosemide (<20% Pills Remaining at Scheduled Pill Counts) at Week 19
Description: Participants' adherence to furosemide will be assessed at scheduled pill counts conducted by the study team at study week 19. Participants' adherence to furosemide will be defined <20% pills remaining at the scheduled pill counts. The percentage of participants who are adherent to furosemide will be determined.
Time Frame: Study week 19 (19 weeks after study medication start)
Population: 23 participants completed the week 19 pill counts. Thus, the analysis population is 23 participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Study Drug Administration: Furosemide
Number analyzed (Participants) | 23
Percentage of participants | 70

ADVERSE EVENTS:
Time Frame: From the time informed consent was obtained to study participation end (up to 24 weeks).
Description: All participants received oral furosemide. Per protocol, adverse events were collected irrespective of dose received and were summarized as a single arm. Of those participants reporting severe or very severe patient-reported outcomes, only severe tinnitus and hearing change were study-defined adverse events per the study protocol.
Groups:
- Study Drug Administration: Furosemide: Open label dose escalation study of furosemide in people receiving maintenance hemodialysis. Participants will take furosemide oral tablets twice daily for 18 weeks. This was a single-arm study with 2 periods. Period 1 is the dose escalation phase. During period 1 (first 6 weeks), the drug dose will be escalated every 2 weeks if safe, tolerated, and acceptable to the participant. Period 2 is the follow-up phase. During period 2 (subsequent 12 weeks), all participants will take the maximum tolerated dose from study period 1, received every 4 weeks if safe, tolerated, and acceptable to the participant.
  First 2 weeks of the study: participants not taking oral furosemide at enrollment will take 80mg furosemide twice daily, those taking oral furosemide at enrollment will stay on their prescribed dose, and those taking another loop diuretic at enrollment will discontinue their prescription and take an equivalent oral furosemide dose. At week 4: dose escalation if tolerated (from 80mg to 120mg twice daily for the 1st group, and a 50% increased dose not >320mg/day for the 2nd & 3rd groups). At week 6: dose escalation if tolerated (from 120mg to 160mg twice daily for the 1st group, and a 50% increased dose not >320mg/day for the 2nd & 3rd groups). Final 12 weeks: all participants will take the maximum tolerated dose (period 2).
  All participants received oral furosemide. Per protocol, adverse events were collected irrespective of dose received and were summarized as a single arm.
Arm/Group | Study Drug Administration: Furosemide
All-Cause Mortality (participants affected / at risk) | 2/39
Serious Adverse Events (participants affected / at risk) | 8/39
Other Adverse Events (participants affected / at risk) | 6/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug Administration: Furosemide (N=39)
Hospitalization for stroke (Nervous system disorders) | 1 (1)
Hospitalization for cardiogenic shock (Cardiac disorders) | 1 (1)
Hospitalization for clostridium difficile infection (Infections and infestations) | 1 (1)
Hospitalization for COVID-19 infection (Infections and infestations) | 2 (2)
Death due to COVID-19-related respiratory failure (Infections and infestations) | 1 (1)
Hospitalization for acute respiratory failure due to volume overload (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for non-ST-elevation myocardial infarction (Cardiac disorders) | 1 (1)
Hospitalization for toe osteomyelitis requiring amputation (Surgical and medical procedures) | 1 (1)
Hospitalization for perforated ulcer, resulting in patient death (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug Administration: Furosemide (N=39)
Inner EAR hearing assessment score decreased by >10 points from baseline (Ear and labyrinth disorders) | 3 (4)
Hypotension during dialysis treatment (Renal and urinary disorders) | 2 (2)
Severe tinnitus (Ear and labyrinth disorders) | 1 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT04622709/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT04622709/ICF_001.pdf